CLINICAL TRIAL: NCT06715527
Title: Treatment of Women With Different Phenotype of Polycystic Ovary Syndrome
Brief Title: Treatment of Women With Hyperandrogenic PCOS With Two Different Ratios of Myo-inositol:D-chiro-inositol: A Comparison
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lo.Li.Pharma s.r.l (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ino-ratio_2024
Record Dates: First submitted 2024-11-28; First posted 2024-12-04 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Polycystic Ovarian Syndrome (PCOS)
Keywords: PCOS; myo-inositol; D-chiro-inositol; menstual cycle
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Inositol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Experimental): Women with PCOS under oral supplementation with myo-inositol and D-chiro-inositol in 40:1 ratio
  Interventions: Dietary Supplement: Myo-Inositol and D-Chiro-Inositol (40:1)
- Comparator (Active Comparator): Women with PCOS under oral supplementation with myo-inositol and D-chiro-inositol in 3.6:1 ratio
  Interventions: Dietary Supplement: Myo-Inositol and D-Chiro-Inositol (3.6:1)

INTERVENTIONS:
Dietary Supplement: Myo-Inositol and D-Chiro-Inositol (40:1) — Myo-inositol and D-chiro-inositol (40:1 ratio), 2 grams (twice a day) for three months
  Other Names: 40:1
  Arms: Treatment
Dietary Supplement: Myo-Inositol and D-Chiro-Inositol (3.6:1) — Myo-inositol and D-chiro-inositol (3.6:1 ratio), 1.4 grams (once daily) for three months
  Other Names: 3.6:1
  Arms: Comparator

SUMMARY:
In this study, female patients diagnosed with polycystic ovary syndrome (PCOS) will be enrolled. In particular, those with elevated testosterone or with clinical signs of hyperandrogenism, along with menstrual cycle alterations and/or polycystic ovary morphology at ultrasound, will be included in the study.

Current treatments for PCOS include insulin sensitizers (such as metformin) and hormonal contraceptives. However, they are not devoid of side effects or may not be well tolerated, often leading to therapy discontinuation. Inositol represents a valid alternative to standard treatments, as it serves both as insulin sensitizer and as second messenger of FSH in the ovaries, thus regulating glucose metabolism and supporting ovarian function. The presence of two inositol isomers, namely myo-inositol and D-chiro-inositol, in defined ratios in human tissues suggests that supplementation with both would be ideal. Despite numerous evidence available, the ratio that gives the best clinical results is still debated.

In the present clinical trial, patients will be given a dietary supplement containing myo-inositol and D-chiro-inositol in two ratios (either 40:1 or 3.6:1, respectively) for three months. Restoration of regular menstrual cycle and of hormonal status will be the primary goal of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* PCOS according to the Rotterdam Criteria
* Clinical or biochemical hyperandrogenism

Exclusion Criteria:

* other causes of ovulatory disfunction (e.g., hyperprolactinemia or hypothyroidism)
* other causes of hyperandrogenism (e.g., adrenal hyperplasia or Cushing's syndrome)
* use of medications that influence ovulation
* hormonal treatments
* chronic pharmacological therapies
* use of inositol-containing supplements
* regular consumption of inositol-enriched food

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-03-06 (Actual); Study Completion 2025-03-14 (Actual)

PRIMARY OUTCOMES:
Restoration of regular menstrual cycle | From enrollment (T0) to the completion of the study at 3 months (T3M)
  Number (%) of patients with regular menstrual cycle at the end of the study

SECONDARY OUTCOMES:
Hormonal status | From enrollment (T0) to the completion of the study at 3 months (T3M)
  Changes of serum hormonal levels (Progesterone; FSH; LH; Estradiol; Testosterone; Insulin)

CONTACTS AND LOCATIONS:
Locations (1):
- Alma Res Fertility Center, Rome, ITA, Italy

IPD SHARING:
Plan to Share IPD: No